CLINICAL TRIAL: NCT06840132
Title: The Effect of Ankle Foot Orthesis on Task-oriented Treatment in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Collaborators: Balikesir Ataturk City Hospital (Other Government)
Responsible Party: Principal Investigator, Sezen Dincer, assistant professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Balıkesir Atatürk CityHospital
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: stroke; foot orthoses; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Exercise; Orthotic Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the task-oriented training (Active Comparator): patients participated in an intensive physical therapy program for 1 hour per day, 5 days a week, over a period of 4 weeks. For GoPT, a 7-station exercise protocol was designed, consisting of motor activities progressing from easy to difficult, with the goal of transforming these activities into permanent skills through meaningful tasks. Each station aimed to gradually improve the patient's motor abilities. Patients were allowed to rest between tasks, and the difficulty of the tasks progressively increased based on each patient's capacity. This 7-station protocol was designed for the first time by our own research team, and the details of the GoPT program
  Interventions: Procedure: Exercise
- the task-oriented training plus plastic static ankle-foot orthosis group (Active Comparator): patients participated in an intensive physical therapy program for 1 hour per day, 5 days a week, over a period of 4 weeks. group using plastic static ankle-foot orthoses (GoPT+AFO) performed the same 7-station exercise protocol as the GoPT group. However, participants in this group were required to wear custom-made plastic static ankle-foot orthoses while completing the exercises. Both the patients and their families were educated on the proper use of the orthosis and encouraged to wear it in daily life as well.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — 7-station exercise protocol was designed, consisting of motor activities progressing from easy to difficult, with the goal of transforming these activities into permanent skills through meaningful tasks. Each station aimed to gradually improve the patient's motor abilities. Patients were allowed to rest between tasks, and the difficulty of the tasks progressively increased based on each patient's capacity. This 7-station protocol was designed for the first time by our own research team
  Other Names: task oriented exercise therapy
  Arms: the task-oriented training
Procedure: Exercise — In addition to the task-oriented training program, the group using plastic static ankle-foot orthoses performed the same 7-station exercise protocol as the task oriented training group. However, participants in this group were required to wear custom-made plastic static ankle-foot orthoses while completing the exercises.
  Other Names: task oriented training + orthoses
  Arms: the task-oriented training plus plastic static ankle-foot orthosis group

SUMMARY:
A stroke is a neurological condition and a major cause of disability in adults. It occurs suddenly and causes specific brain function problems, leading to noticeable symptoms that last for more than 24 hours.Stroke commonly causes impairments in sensory, motor, and cognitive functions. Approximately 80% of patients experience motor deficits in the lower extremities, often accompanied by balance disturbance (3). Traditionally, neurodevelopmental treatments aimed at restoring normal movement patterns have been used in stroke rehabilitation. However, research on both animals and humans has shown that this approach alone is insufficient. These studies have shown that task-oriented functional exercise training can induce changes in activation patterns in a large portion of the damaged brain areas, leading to restoration of function (4, 5). Engaging in meaningful and repetitive goal-directed functional tasks can effectively enhance neuroplasticity and facilitate recovery.

Task-oriented training is an exercise therapy designed for stroke patients, based on motor learning theory, which emphasizes the repetition of motor skills and aims to enhance performance through meaningful tasks . Lord et al. were the first researchers to conceptually apply task-oriented training, using a total of 19 different functional exercises in their study. They found that both deficiency-based and task-oriented training showed similar results in terms of improving walking and balance skills. However, more recent studies have shown that task-specific, task-oriented treatment programs are superior to traditional facilitation-based therapeutic approaches. Another study comparing conventional physiotherapy, task-oriented group training, and individual task-oriented training, with the aim of assessing the effects of exercises, demonstrated that task-oriented group training led to better outcomes in tasks such as sitting, standing, overcoming obstacles, circular walking, and carrying objects.

Two others found that the foot was more dorsiflexed at higher stiffnesses during initial contact in patients post- stroke An Ankle-Foot Orthosis (AFO) plays a crucial role in individuals with paralysis during walking, particularly in the heel strike and loading phases, by restraining plantar flexion and assisting the impaired function of the dorsiflexors. In individuals with paralysis, dorsiflexion, the upward movement of the ankle, is often weakened or lost. The AFO helps address this issue by maintaining the desired position of the ankle joint, contributing to the preservation of normal gait during walking.

Additionally, during the swing phase (when the leg moves forward), the AFO helps maintain the ankle joint position, supporting toe-off. This enhances walking efficiency and provides stability during the step. Thus, the AFO not only offers support but also significantly contributes to functional improvement, greatly enhancing the walking ability of individuals with paralysis.

Combined use of task-oriented training and orthoses are typically focused on the upper extremity functions rather than the lower extremity functions in patients with stroke. Therefore, in this study, it was aimed to investigate the effects of task-oriented training with and without an ankle-foot orthosis (AFO) on lower extremity function in individuals with stroke. It was hypothesized that task-oriented training with an AFO would lead to greater improvements in lower extremity function such as balance, walking, and stability and quality of life in stroke patients.

The study included 40 individuals with stroke. The inclusion criteria of the study were as follows: aged 18 and older, who had experienced their first stroke, Brunnstrom lower extremity score of ≥3, a Functional Ambulation Classification score of ≥2, at least 3 months post-stroke, and having no other neurological disorders. The individuals will be diagnosed at the Physical Therapy and Rehabilitation outpatient clinic of Balıkesir Atatürk City Hospital by the same neurologist and received treatment at the hospital's rehabilitation department.All patients participated in an intensive physical therapy program for 1 hour per day, 5 days a week, over a period of 4 weeks. For GoPT, a 7-station exercise protocol designed, consisting of motor activities progressing from easy to difficult, with the goal of transforming these activities into permanent skills through meaningful tasks. Participants randomly divided into two groups: the task-oriented physical therapy group (GoPT) (n=19), the task-oriented program plus plastic static ankle-foot orthosis group (GoPT+AFO) (n=20). All participants in the groups were evaluated by a physiotherapist before treatment and after the 4-week intervention period.Six-Minute Walk Test, 10-Meter Walk Test,Timed Up and Go Test,Berg Balance Scale, Functional Reach Test,Stroke Impact Scale were evaluated.

DETAILED DESCRIPTION:
Before starting the study, an application was made to Balıkesir University Non-Interventional Clinical Research Ethics Committee. Usage started with the permission of the ethics committee, decision dated 13.12.2017 and 2017/156.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older,
* Who had experienced their first stroke,
* Brunnstrom lower extremity score of ≥3,
* Functional Ambulation Classification score of ≥2,
* At least 3 months post-stroke,
* Having no other neurological disorders

Exclusion Criteria:

* Under 18 age,
* Having an another neurologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
six meter walk | from enrollement to the end of four weeks
  endurance test. It is assessed by having the person walk continuously for 6 minutes at the maximum speed they can walk in a 30-meter area. The distance walked during this time is recorded. Increased walking distance is perceived positively

SECONDARY OUTCOMES:
berg balance scale | from enrollement to the end of 4 weeks
  balance evaluation. Each activity is given a score between 0-4. The best score is 56. 0-20 is interpreted as poor balance, 21-40 as acceptable balance, and 41-56 as advanced balance skills.

CONTACTS AND LOCATIONS:
Overall Officials: sezen dincer, asst prof, Principal Investigator — ankara medipol univercity
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Song HS, Kim JY, Park SD. The effect of class-based task-oriented circuit training on the self-satisfaction of patients with chronic stroke. J Phys Ther Sci. 2015 Jan;27(1):127-9. doi: 10.1589/jpts.27.127. Epub 2015 Jan 9. PMID 25642055
- [Result] French B, Thomas LH, Coupe J, McMahon NE, Connell L, Harrison J, Sutton CJ, Tishkovskaya S, Watkins CL. Repetitive task training for improving functional ability after stroke. Cochrane Database Syst Rev. 2016 Nov 14;11(11):CD006073. doi: 10.1002/14651858.CD006073.pub3. PMID 27841442
- [Result] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848